CLINICAL TRIAL: NCT04197947
Title: Selectively Modulating Pathophysiological Biomaker to Improve Freezing of Gait in Parkinson' s Disease by Adaptive Subthalamic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802209A0
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-02

CONDITIONS: Freezing of Gait; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD patient who have FoG (Experimental)
  Interventions: Device: Neuro Omega

INTERVENTIONS:
Device: Neuro Omega — A neurophysiological navigation system NeuroOmegaTM (Alpha Omega. Israel) was implemented in our group and the operation of this system for aDBS experiment is proved to be successful (Fig 9, 10). This system was proved by both FDA and tFDA. The aDBS stimulation algorithm will be integrated with NeuroOmegaTM. The aDBS stimulation control will achieve through self-developed algorithms or built-in scripting of the system. We introduce NeuroOmega system to conduct the designed aDBS experiment for its multifunction and safety. Our group has established collaboration with Department of Eelectronic Engineering in Chang Gung University (Co-PI HL Chan) and BERTEC in National Ciao Tung University (Co-PI MD Ker). Three postdoctor fellows and one senior engineer have been working on the operation of this aDBS system.
  All hardware and software problems could be sorted out in time.

SUMMARY:
Freezing of gait (FoG) is defined as a brief, episodic absence or reduction of forward progression of the feet despite the intention to walk. It is one of the most disabling and intractable motor symptoms in patients with Parkinson's disease (PD) as it often causes falls and loss of independence. The pathophysiology of FoG remains unclear but it seems differ from other cardinal motor symptoms in PD. The therapeutic efficacy of medical and surgical treatments for FoG are usually suboptimal. Deep brain stimulation (DBS) in the subthalamic nucleus (STN) is a well established treatment for advanced PD with motor fluctuation. It alleviates tremor, bradykinesia and rigidity and improved the quality of life. However, the therapeutic effects of DBS are impeded by high cost of device, stimulation induced adverse effects and partial treatment for some parkinsonism symptoms, particular gait disturbance and FoG. Recently, a new mode of stimulation is proposed. Differing from the conventional DBS which is operated in open loop so that stimulation remains fixed over time and is delivered at regular and high frequencies, the new adaptive DBS (aDBS) detects the pathological activities and only deliver stimulation when it is necessary. Recent studies in MPTP-primate and patients with PD demonstrate that the aDBS is superior to standard continuous DBS. However, the therapeutic efficacy is only shown in "appendicular symptoms" such as bradykinesia, rigidity and tremor. There is no report about the effect of aDBS on gait disturbance, particular FoG in PD so far.

The aim of the current project is to test whether the therapeutic efficacy of aDBS is superior to conventional DBS in PD patients with FoG. To this end, 20 advanced PD patients who undergo STN DBS implantation for the treatment of their disorders will be examined. The gait of patients will be assessed during conventional open loop stimulation and aDBS and the therapeutic efficacy for FoG will be defined. The results of this study will also contribute to better understanding of pathophysiology of FoG and to future development of embedded aDBS system for PD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age between 20 and 75 years old
2. Idiopathic PD with cardinal motor impairment (bradykinesia, rigidity, tremor and postural instability
3. Advanced PD as determined by Hoehn and Yahr stage or UPDRS part III motor score
4. Levodopa responsive
5. Disabling Parkinson's symptoms or drug side effects (dyskinesia, motor fluctuation or disabling "off"period) despite the best medical therapy.
6. Willingness and ability to cooperate during conscious operative and experimental procedure.
7. Normal MRI

Exclusion Criteria:

1. Non-idiopathic parkinsonism or "Parkinson's plus syndrome"
2. Impaired cognitive dysfunction (MMSE<26)
3. Moderate to severe depression (BDI≧30)
4. Depression (BDI≧30), or psychiatric disorder
5. Structure lesion such as stroke, tumor or severe brain atrophy revealed by MRI
6. Major medical disorders, such as hematological, heart disease or malignancy
7. Significant medical, surgical or neurological co-morbidities contraindicating DBS surgery or stimulation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-01-23 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 1 year
  The total motor score of UPDRS (UPDRS III) will be assessed. The subscore of UPDRS item 14 (FoG score) will be test.
Questionnaire of FoG (FoG-Q) | 1 year
  FoG is difficult to measure due to its unpredictable occurrence. FoG-Q was validated in a large, prospective interventional study for the assessment of FoG severity in PD. In addition, it was found to be a reliable tool for assessment of treatment intervention.
Quantitative evaluation of FoG | 1 year
  Patients will be asked to walk at their preferred speed along a path 10 m long for 5 times. A triaxial accelerometer (ACC) (TMSI) will be fixed with tape over spinous processes at the upper thoracic level to record trunk acceleration. The episode of FoG will be recorded by both video and the results of Acc signals.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan District, Taiwan